CLINICAL TRIAL: NCT00763477
Title: The Effect of Ghrelin on Appetite and Immune Function in Patients With Cystic Fibrosis
Brief Title: Ghrelin in Cystic Fibrosis
Acronym: ghrelin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Dr. Alistair Grant, Papworth Hospital NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: P01276
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Weight; Appetite; Ghrelin; Cystic fibrosis with low BMI
MeSH Terms: conditions — Cystic Fibrosis; Body Weight | interventions — Ghrelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- saline injections (Placebo Comparator)
  Interventions: Biological: ghrelin

INTERVENTIONS:
Biological: ghrelin — subcutaneous injection

SUMMARY:
Background to ghrelin Ghrelin is a naturally occurring hormone found in the blood which stimulates appetite. In healthy individuals, levels of ghrelin are high before a meal and falls afterwards. Previous studies have shown that giving ghrelin (by injection) to thin patients with renal failure and cancer increases their food intake. Furthermore, addition of ghrelin may also reduce inflammation within the body. Cystic Fibrosis (CF) is a genetic disease which frequently results in recurrent lung infections (leading to progressive inflammatory lung damage) and low body weight. Low body weight in CF is associated with increased lung infections, rapidly worsening lung function and a shortened life expectancy.

The researchers postulate that administration of extra ghrelin to CF patients with low body weight may increase food intake and reduce lung inflammation. If successful, this study might identify ghrelin as a potential therapy for CF patients to improve nutrition, decrease lung inflammation and thereby improve survival.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the role of a naturally occuring hormone called ghrelin on appetite, energy expenditure and immune function in patients with cystic fibrosis.

Theoretical framework:

Despite advances in the molecular understanding of the disease, life-expectancy in Cystic Fibrosis (CF) remains severely limited. Reduced body-weight is associated with increased inflammatory lung damage and is a major predictor of mortality in CF patients. Malnutrition is highly prevalent in the CF population and results from both poor food intake and excessive energy expenditure. A therapy which improves nutrition may therefore have a significant effect on the prognosis of this disease. Ghrelin is the only physiological circulating factor that is known to increase food intake. Administration of acylated ghrelin to humans increases both hunger and food intake and has been found to increase appetite in chronic disease states associated with anorexia and weight loss (such as cancer and chronic renal disease). From multiple animal and in vitro human studies, ghrelin also appears to have anti-inflammatory properties which would potentially benefit CF patients in whom a chronic inflammatory state promotes lung destruction, malnutrition and increases mortality. Ghrelin replacement may therefore improve nutrition and decrease the inflammatory burden in CF patients, leading to an improvement in life-expectancy. If ghrelin is identified as having an important pathophysiological role in CF it may lead to a future study of its efficacy as a therapeutic agent.

Design Methodology: The study has three sections:

1. a cross sectional study of the levels of blood metabolic signals in participants with cystic fibrosis and healthy controls.
2. a laboratory study of the effect of ghrelin on immune cells extracted from the blood of participants with cystic fibrosis and healthy controls
3. a cross-over interventional study of repeated ghrelin administration in malnourished cystic fibrosis patients

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis
* BMI </=19 kg/m2

Exclusion Criteria:

* Needle phobia
* Pulmonary infection requiring intravenous antibiotics in the past 2 weeks-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-02 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Appetite | 4 weeks

SECONDARY OUTCOMES:
weight | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Papworth Hospital NHs Foundation Trust, Cambridge, Cambridgeshire, United Kingdom